CLINICAL TRIAL: NCT04847258
Title: Rate of Non-copers to Non-surgical ACL Treatment After 3 Months of Rehabilitation - a Prospective Cohort Study
Brief Title: Rate of Non-copers to Non-surgical ACL Treatment After 3 Months of Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ACL screening
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard rehabilitation — Patients follow standard municipal rehabilitation

SUMMARY:
The aim is to determine the sensitivity and specificity of a screening tool to identify patients who undergo ACL reconstruction (non-copers) after 3 months of standard rehabilitation following an anterior Cruciate ligament (ACL) injury.

DETAILED DESCRIPTION:
All included patients are referred to municipal rehabilitation to resolve effusion and range of motion deficits before the first screening (baseline screening) is completed. Hereafter the patients follow 3 months municipal rehabilitation before the second screening (3 months screening). A physiotherapist performs the screening and at the second screening, this is performed prior to consulting an orthopaedic surgeon.

ELIGIBILITY:
Inclusion Criteria:

* unilateral primary ACL injury
* Index injury no older than 6 months

Exclusion Criteria:

* Multiligament rupture
* Large cartillage or meniscus injuries
* Scheduled ACL reconstruction within 3 months

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the outpatient clinic at the Department of Orthopaedic Surgery at Vejle Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 357 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients undergoing ACL reconstruction after 3 months of standard rehabilitation | 3 months
  Patients undergoing ACL reconstruction after 3 months of standard rehabilitation are defined as non-copers to the non-surgical treatment, which will define the sensitivity and specificity of the screening examination.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Varnum, ph.d., Study Director — Vejle Hosptal
Locations (1):
- Vejle Hospital, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided